CLINICAL TRIAL: NCT05892653
Title: A Phase I, Open-Label, Multicenter Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics &Preliminary Anti-Cancer Efficacy of ABM-1310 in Patients With BRAF V600-Mutant Relapsed &Drug Resistant Primary Malignant Brain Tumors
Brief Title: A Study of ABM-1310 in Patients With BRAF V600-Mutant Relapsed and Drug Resistant Primary Malignant Brain Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Adjustment of the applicant's research and development strategy
Sponsor: ABM Therapeutics Shanghai Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABM1310X1102C
Record Dates: First submitted 2023-05-18; First posted 2023-06-07 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Primary Malignant Brain Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose Escalation and Dose Expansion (Experimental): During the dose escalation stage, a classic "3+3" design will be used to guide dose escalation to determine MTD and RP2D. Three to six subjects are expected to be enrolled in each dose group and at least 6 subjects are enrolled in the MTD/highest dose group. The total number of subjects enrolled during the dose escalation stage will depend on the amount of DLT and the total number of dose levels explored. If DLT is not observed in the first 3 subjects enrolled for each dose level, the Safety Monitoring Committee (SMC) will review the cumulative safety data of subjects at each dose level and decide whether to proceed with dose escalation upon the completion of study treatment at least for the DLT evaluation period (28 days of Cycle 1). The dose expansion stage in this study will be initiated at the MTD or the optimal dose determined by the SMC as a fixed dose level (MTD or the optimal dose needs to be reviewed by the SMC and subjects are safe and tolerable at that dose level).
  Interventions: Drug: ABM-1310

INTERVENTIONS:
Drug: ABM-1310 — Dose Escalation Stage: Subjects will be given oral dosing of ABM-1310 twice daily (BID) for 28-day cycles of continuous administration until progressive disease (PD), unacceptable toxicity, or other withdrawal criteria are met as clinically observed.
  Dose Expansion Stage: Subjects will begin to receive oral doses of ABM-1310, BID, for 28-day cycles at a fixed dose level (as determined at the dose escalation stage) until PD, unacceptable toxicity, or other withdrawal criteria are met as clinically observed.

SUMMARY:
Overall Design: This is a phase I, open-label, multicenter clinical study to evaluate the safety, tolerability, pharmacokinetics, and preliminary anti-cancer efficacy of ABM-1310 in patients with BRAF V600-mutant relapsed and drug resistant primary malignant brain tumors.

The study including four periods of screening (28 days), treatment (no more than 2 years), safety follow-up and survival follow-up.

This study consists of two stages: dose escalation and dose expansion. During the dose escalation stage, a classic "3+3" design will be used to guide dose escalation to determine MTD and RP2D. Three to six subjects are expected to be enrolled in each dose group and at least 6 subjects are enrolled in the MTD/highest dose group. The total number of subjects enrolled during the dose escalation stage will depend on the amount of DLT and the total number of dose levels explored. If DLT is not observed in the first 3 subjects enrolled for each dose level, the Safety Monitoring Committee (SMC, including investigators, pharmacologists, and the sponsor's medical specialists, and other experienced members specially invited as necessary) will review the cumulative safety data of subjects at each dose level and decide whether to proceed with dose escalation upon the completion of study treatment at least for the DLT evaluation period (28 days of Cycle 1).

The dose expansion stage in this study will be initiated at the MTD or the optimal dose determined by the SMC as a fixed dose level (MTD or the optimal dose needs to be reviewed by the SMC and subjects are safe and tolerable at that dose level). The dose expansion stage is expected to include the following two cohorts of relapsed and drug resistant primary malignant brain tumors with BRAF V600 mutations:Cohort 1: GBM, N = up to 25 patients; Cohort 2: In addition to GBM, other primary malignant brain tumors, N = up to 15 patients.

In this study, the corresponding sample size for each cohort/tumor type may be determined according to the actual efficacy and safety data obtained. After each cohort included the first 10 patients, the available safety, efficacy, and PK data were analyzed. Based on the analysis results, the sponsor decided whether to continue recruiting patients for the study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are able to understand and voluntarily sign informed consent forms (ICFs).
2. Male and female subjects at the age of ≥18 at the time of screening.
3. Patients with histologically or cytologically-confirmed, primary malignant brain tumor with (a) failure of prior standard therapy, (b) no standard therapy available, or (c) for whom standard therapy is not applicable considered by the patient or treating physician, or (d) intolerance to standard treatment. Subjects who were previously treated with BRAF and/or MEK inhibitors are allowed to be enrolled in this study.
4. Documentation of positive BRAF V600 mutation is required for enrollment. It is recommended to provide sufficient fresh/archived tumor tissue samples (formalin-fixed paraffin-embedded tumor specimens [preferred]) or 5-10 available unstained sections of good quality for verification of BRAF V600 mutation status at the central laboratory. For any subject who is unable to provide suitable and adequate tumor specimens, re-biopsy (with controllable safety) can be performed in a non-mandatory manner if it is feasible as assessed by the investigator and the subject gives informed consent; if re-biopsy is impossible or refused by the subject, his/her eligibility for enrollment shall be confirmed by both the investigator and the sponsor.
5. Patients with primary malignant brain tumors that are asymptomatic, or that are symptomatic but on a stable or decreasing dose of steroids for at least 2 weeks are eligible for enrollment. The specific criteria are as follows:Subjects with inactive and asymptomatic primary malignant brain tumors;Subjects who have active, mild neurological signs and symptoms currently requiring no therapy with steroids, and have no history of epileptic seizure within 2 weeks prior to initiation of treatment;Subjects who have active, neurological signs and symptoms and were on a stable or gradually reducing dose up to 5 mg of dexamethasone (or equivalent) per day within 2 weeks prior to initiation of treatment;
6. Antitumor efficacy was evaluated using the RANO criteria, which required the presence of at least one measurable lesion (the diameters that are perpendicular to each other are not less than 10 mm). Lesions previously treated with radiotherapy shall not be deemed as target lesions unless significant progression as shown on imaging.
7. Karnofsky PS score of ≥ 60.
8. Survival expectancy ≥ 3 months.
9. Adequate organ function (no blood transfusion and no use of granulocyte colony-stimulating factor, or other hematopoietic stimulator support within 2 weeks before the first administration of the study drug) confirmed as evidenced by:Absolute Neutrophil Count (ANC) ≥ 1.5×10^9/L;Hemoglobin (Hgb) ≥ 90 g/dl;Platelets (Plt) ≥ 75×10^9/L;AST/ALT ≤ 2.5 x ULN or ≤ 5.0 x ULN if liver metastases are present;Bilirubin total ≤ 1.5 x ULN, or bilirubin direct < ULN for patients with bilirubin total levels >1.5 ULN;Serum creatinine < 1.5 x ULN or creatinine clearance > 50 mL/min (as calculated via Cockcroft-Gault formula based on the actual body weight of the subject;International normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5 x ULN for subjects not receiving anticoagulant therapy, and INR is maintained within the standard range of treatment prior to starting study drug for subjects receiving anticoagulant therapy.
10. Hepatitis B virus surface antigen (HBsAg) is negative, or HBsAg is positive but HBV DNA titer is below the lower limit of positive detection of the participating site at screening.HBsAg-positive or HBV-DNA positive subjects shall be managed according to institutional guidelines (anti-HBV therapy, where appropriate, and close monitoring of liver function and HBV-DNA replication shall be performed).
11. Negative hepatitis C virus (HCV) antibody test or positive HCV antibody test at the time of screening followed by a negative HCV-RNA test result.HCV-RNA testing is performed only for subjects with a positive HCV antibody test result.
12. Negative HIV test result at the time of screening.
13. All pre-menopausal women and women with menolipsis < 12 months should have a negative pregnancy test result within 7 days before starting study treatment.
14. Must agree to take sufficient contraceptive methods before initiation of study treatment, during the study, and for at least 3 months after the last dose of the study drug.
15. Subjects who are able to swallow a capsule in whole (without chewing, crushing, or opening).

Exclusion Criteria:

1. Women who are pregnant or breast-feeding.
2. Subjects with history of neoplasm malignant (except for primary malignant brain tumors) within 5 years prior to screening, excluding cured carcinoma in situ of cervix, non-melanoma skin cancer, localized prostate cancer and other tumors/cancers that have undergone radical treatment and shown no signs of disease for at least 3 years (This exclusion criterion is only applicable for dose expansion stage). For the dose escalation stage, any patient with double primary malignant solid tumors who can indeed benefit from this study as confirmed by the investigator is eligible for the screening.
3. Subjects with intracranial hypertension or associated risks (e.g., intracranial infection, intracranial hemorrhage) to be controlled.
4. Subjects with clinically uncontrolled pleural effusion, pericardial effusion, or ascites who, in the judgement of the investigator, are not eligible for enrollment.
5. Subjects with history of symptomatic stroke within 6 months prior to initiation of study treatment.
6. Subjects with epileptic seizure within 14 days prior to initiation of study treatment.
7. Impaired cardiac function or clinically significant cardiovascular disorder, including but not limited to any of the following:Left Ventricular Ejection Fraction (LVEF) < 50% as determined via cardiac ultrasound.Long QT syndrome congenital.QTcF (as corrected via Fridericia formula) ≥ 450 ms at screening.Second-degree type II AV block or third-degree AV block.Unstable angina pectoris within 6 months prior to starting study drug.Acute myocardial infarction within 6 months prior to starting study drug.New York Heart Association (NYHA) Class II or higher heart failure within 6 months prior to study treatment.Ventricular arrhythmias > Grade 2 within 6 months prior to study treatment.Poorly controlled hypertension as defined as systolic blood pressure of >160 mmHg or diastolic blood pressure of > 100 mmHg despite use of antihypertensive medications.Combined with any pulmonary embolism, or presence of any serious deep vein thrombosis on lower extremities that require medical interventions such as vena cava filter insertion at the screening.
8. Poorly controlled diabetes (fasting glucose > 10 mmol/L or Glycosylated Haemoglobin (HbA1c) > 8%) despite standard drug therapy.
9. Subjects with:CTCAE grade 2 or higher unresolved diarrhea, or Impaired gastrointestinal (GI) function or GI diseases that may significantly alter the absorption of ABM-1310 (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
10. Previous or current, Grade 2 or higher eye disorder, such as retinal vein occlusion (RVO).
11. Severe chronic or active infections requiring intravenous anti-infective therapy within 2 weeks prior to study treatment, including but not limited infectious complications leading to hospitalization, bacteremia, severe pneumonia, or active tuberculosis.Subjects with local fungal infections of skin or nails are allowed for enrollment. Subjects receiving prophylactic antibiotics (e.g., to prevent urinary tract infections or exacerbations of chronic obstructive pulmonary disease) are eligible for study (except for antibiotics prohibited by the protocol).
12. Subjects with solid organ or hematopoietic stem cell transplant within the past 5 years.
13. Patients receiving chemotherapy, targeted therapy, or immunotherapy within 4 weeks prior to study treatment, including the followings:Receiving nitrosourea or mitomycin-C within 6 weeks prior to study treatment.Receiving fluorouracil or small molecule targeted drug therapy within 5 half-lives or 2 weeks (whichever is longer) prior to study treatment.Receiving Chinese herbal or patent medicine within 2 weeks prior to study treatment for anti-tumor indications.
14. Patients receiving radiotherapy to head within 4 weeks prior to study treatment.
15. Adverse reactions resulted from prior antitumor therapy that have not resolved to baseline or ≤ grade 1 (CTCAE 5.0) , except alopecia or ≤ grade 2 peripheral neuropathy, hypothyroidism stabilized by hormone replacement therapy, etc.
16. Subjects who have undergone major surgery within 4 weeks prior to study treatment or who have not recovered from side effects of such therapy or who are expected to undergo major surgery during study treatment. However, a minimum of 2 weeks recovery time from major surgery to starting study drug is required if in investigator's opinion the patient has recovered from such major surgery.
17. Subjects currently receiving therapeutic doses of warfarin sodium or any other coumarin-derivative anticoagulants.
18. Subjects who are currently receiving treatment with medication that has a known risk to prolong the QT interval and cannot either be discontinued or switched to a different medication prior to starting study drug.
19. Known, documented or suspected history of drug abuse, expect opioids prescribed for pain relief, etc.
20. Past or current evidence of any condition, therapy, or laboratory abnormality that, in the opinion of the investigator, might affect the results of the study, and interfere with the subject's participation and study compliance.
21. Other severe and/or uncontrolled concomitant diseases that could cause unacceptable safety risks or compromise compliance with the study protocol.
22. Other conditions that, in the judgement of the investigator, are inappropriate for enrollment in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-06-30 (Actual); Primary Completion 2024-08-27 (Actual); Study Completion 2024-08-27 (Actual)

PRIMARY OUTCOMES:
MTD | From the enrollment of subjects to the end of Cycle 1 (each cycle is 28 days) or up to treatment discontinuation, whichever occurs first, assessed up to 28 days.
  MTD is defined as the highest dose level at which DLT is observed in ≤ 1/6 subjects at one single dose group.
Recommended Phase 2 Dose(PR2D) | From the enrollment of subjects to the end of Cycle 1 (each cycle is 28 days) or up to treatment discontinuation, whichever occurs first, assessed up to 28 days.
  RP2D will be a dose either below or equal to MTD
Dose Limiting Toxicity(DLT) | cycle 1（28 days）
  DLT will be evaluated according to NCI-CTCAE V5.0 criteria
The incidence of treatment-related adverse events AE(s) | Up to 28 days from treatment discontinuation
  Safety and tolerability of ABM-1310 monotherapy
Number of participants with abnormal laboratory values | Up to 28 days from treatment discontinuation
  Safety and tolerability of ABM-1310 monotherapy
Number of participants with abnormal vital signs | Up to 28 days from treatment discontinuation
  Safety and tolerability of ABM-1310 monotherapy
Number of participants with abnormal physical examinations | Up to 28 days from treatment discontinuation
  Safety and tolerability of ABM-1310 monotherapy
Number of participants with abnormal ophthalmic evaluation | Up to 28 days from treatment discontinuation
  Safety and tolerability of ABM-1310 monotherapy
Number of participants with abnormal ECG | Up to 28 days from treatment discontinuation
  Safety and tolerability of ABM-1310 monotherapy
Number of participants with abnormal Karnofsky PS | Up to 28 days from treatment discontinuation
  Safety and tolerability of ABM-1310 monotherapy

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | From the enrollment of subjects to the time of disease progression in radiological imaging or death from any cause, whichever occurs first, assessed approximately 12 months.
  Preliminary efficacy of ABM-1310 monotherapy
Disease Control Rate(DCR) | From the enrollment of subjects to the time of disease progression in radiological imaging or death from any cause, whichever occurs first, assessed approximately 12 months.
  Preliminary efficacy of ABM-1310 monotherapy
Duration of Response（DOR） | From the enrollment of subjects to the time of disease progression in radiological imaging or death from any cause, whichever occurs first, assessed approximately 12 months.
  Preliminary efficacy of ABM-1310 monotherapy
Progression free survival (PFS) | From the enrollment of subjects to the time of disease progression in radiological imaging or death from any cause, whichever occurs first, assessed approximately 12 months.
  Preliminary efficacy of ABM-1310 monotherapy
Overall Survival(OS) | From the enrollment of subjects to the time of death from any cause or the study discontinuation, whichever occurs first, assessed approximately 18 months.
  Preliminary efficacy of ABM-1310 monotherapy
Peak Concentration（Cmax） | 12 hours after the first dose on the first day of cycle 1 (each cycle is 28 days)
  Pharmacokinetic (PK) profile of ABM-1310 monotherapy
Time to Cmax(Tmax) | 12 hours after the first dose on the first day of cycle 1 (each cycle is 28 days)
  Pharmacokinetic (PK) profile of ABM-1310 monotherapy
AUC from time 0 to the time of last measurable concentration（AUC0-last) | Up to Day 2, Day 8, Day 15, Day 22 and Day 28 of Cycle 1. Up to Day 1 and Day 2 of Cycle2. After Cycle2, tests every 2 cycles (each cycle is 28 days)
  Pharmacokinetic (PK) profile of ABM-1310 monotherapy
Steady-state Concentration（Css） | At the Day 1 and Day 2 of Cycle 2 (each cycle is 28 days)
  PK characteristics of repeated administration of ABM-1310 monotherapy
Terminal half-life（T1/2） | 12 hours after the first dose on the first day of cycle 1 (each cycle is 28 days)
  Pharmacokinetic (PK) profile of ABM-1310 monotherapy

OTHER OUTCOMES:
Exposure analysis of ABM-1310 in cerebrospinal fluid | At the first day of Cycle 2 (each cycle is 28 days，dose expansion stage only)
  After repeated administration of ABM-1310, the drug exposure of ABM-1310 in cerebrospinal fluid was explored when the blood concentration of ABM-1310 reached stable state.

CONTACTS AND LOCATIONS:
Overall Officials: Wenbin Li, Principal Investigator — Beijing Tiantan Hospital
Locations (4):
- China (4):
  - Beijing Tiantan Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality
  - Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - First affiliated hospital to SuZhou University, Suzhou, Jiangsu
  - Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No